CLINICAL TRIAL: NCT00445835
Title: Active Detection and Management of the Extension of Atherothrombosis in High Risk Coronary Patients In Comparison With Standard of Care for Coronary Atherosclerosis: The AMERICA Study
Brief Title: Active Detection of the Extension of Atherothrombosis in High Risk Coronary Patients
Acronym: AMERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut de l'Atherothrombose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060902; PHAO 2006
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; myocardial infarction; atherothrombosis; atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Thrombosis; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BA :Active arm (Other): A strategy of systematic screening of these extra-coronary asymptomatic lesions combined with a specific treatment if needed and an aggressive secondary prevention pharmacological treatment of atherothrombosis
  Interventions: Other: Arterial doppler for screening asymptomatic and significant extracoronary arterial stenoses in all arterial beds
- BC: Conservative arm (Other): Conservative medical approach
  Interventions: Other: Conservative arm

INTERVENTIONS:
Other: Arterial doppler for screening asymptomatic and significant extracoronary arterial stenoses in all arterial beds — A strategy of systematic screening of these extra-coronary asymptomatic lesions combined with a specific treatment if needed and an aggressive secondary prevention pharmacological treatment of atherothrombosis
  Arms: BA :Active arm
Other: Conservative arm — Conservative medical approach
  Arms: BC: Conservative arm

SUMMARY:
Coronary artery disease is the first cause of death related to atherothrombosis.

DETAILED DESCRIPTION:
Coronary artery disease is the first cause of death related to atherothrombosis. There is a close correlation between the extension of coronary artery disease and the severity of atherosclerotic lesions in extra coronary arterial beds. In addition, these symptomatic extracoronary lesions dramatically decrease the survival of these patients. However, scant data are available regarding the prevalence of extracoronary asymptomatic lesions. Conversely, the annual absolute risk of these lesions remains unknown. Consequently, whether a systematic identification of these extracoronary asymptomatic lesions is relevant remains to be established. The Primary Objective and Primary Endpoint of the AMERICA study is to demonstrate the superiority of an active detection and management of the extension of atherothrombosis in high Risk coronary patients (active strategy) in comparison with standard of care for coronary atherosclerosis (conservative strategy).

ELIGIBILITY:
Inclusion criteria:

1. Three vessel disease recently identified recently (<6 month)
2. Accrue coronary syndromes in patients>75 years old (<1 month)

Exclusion criteria:

1. Absence of significant coronary lesions
2. Other causes of rise in the troponin level
3. Patient<18 years old
4. Pregnant women
5. Patient without affiliation to National Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
death (all cause) or any ischemic event leading to rehospitalisation or any evidence of organ failure. | during the study
  death (all cause) or any ischemic event leading to rehospitalisation or any evidence of organ failure.

SECONDARY OUTCOMES:
Incidence of each composite of the primary endpoint. | during the study
  Incidence of each composite of the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe COLLET, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Pitie-Salpetriere, Paris, France

REFERENCES:
- [Derived] Collet JP, Cayla G, Ennezat PV, Leclercq F, Cuisset T, Elhadad S, Henry P, Belle L, Cohen A, Silvain J, Barthelemy O, Beygui F, Diallo A, Vicaut E, Montalescot G; AMERICA Investigators. Systematic detection of polyvascular disease combined with aggressive secondary prevention in patients presenting with severe coronary artery disease: The randomized AMERICA Study. Int J Cardiol. 2018 Mar 1;254:36-42. doi: 10.1016/j.ijcard.2017.11.081. Epub 2018 Jan 28. PMID 29407124